CLINICAL TRIAL: NCT02987517
Title: A Prospective Study of Interventions Aimed at Reducing Impact Loads in Runners
Brief Title: A Comparative Effectiveness Study of Two Interventions Aimed at Reducing Impact Loads in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Irene Sprague Davis, Director, Spaulding National Running Center, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015P000724
Record Dates: First submitted 2016-12-05; First posted 2016-12-09 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Musculoskeletal Injury
Keywords: running; vertical load rates; cadence; footstrike

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cadence (Experimental): Runners who use an increased running cadence of 7.5 percent over preferred running cadence.
  Interventions: Other: Increased running cadence gait retraining; Other: Strengthening exercises
- Forefoot Strike (Experimental): Runners who use a forefoot strike instead of a rear foot strike
  Interventions: Other: Forefoot Strike gait retraining; Other: Strengthening exercises

INTERVENTIONS:
Other: Increased running cadence gait retraining — Runners use an increased cadence, or step rate, 7.5% greater than baseline preferred cadence
  Arms: Cadence
Other: Forefoot Strike gait retraining — Runners use a forefoot strike running gait instead of a rear foot strike running gait.
  Arms: Forefoot Strike
Other: Strengthening exercises — foot and ankle strengthening exercises performed by all subjects to prepare musculoskeletal tissues for requirements of new running gait.

SUMMARY:
This study will use a comparative effectiveness design of two interventions known to reduce running impacts. The study will be conducted at the Spaulding National Running Center. A total of 40 male and female participants, between ages 18-50 years, running 10- 30 miles per week will be recruited from the local running community. All potential subjects will be cleared for physical activity using a Physical Activity Readiness Questionnaire (PAR-Q) and screened via high-speed video to determine their habitual footstrike pattern. Those who are rearfoot strikers will be included and will then be randomized to either an increased cadence (CAD) or a forefoot strike (FFS) intervention group. Standardized running shoes will be provided to both groups for the duration of the study. All participants will attend 2 strength-training instruction sessions with a physical therapist prior to gait-retraining intervention. They will be instructed to perform the learned exercises daily for 4 weeks to prepare the body tissues for forces associated with new gait methods. Subjects will then attend 8 gait-retraining sessions over 2-3 weeks. Sessions will be scheduled as two sequential days of training followed by a day of rest. The gait retraining protocols will be conducted on a treadmill. 3D Motion Capture analysis will be conducted at baseline and at 3 points following intervention (1 week, 1 month, and 6 months).

DETAILED DESCRIPTION:
SUBJECT ENROLLMENT

When potential participants are contacted (or contact investigators), they will be screened by phone or email to ensure they meet the study inclusion or exclusion criteria. If they do, details of the study procedures will be explained and they will be given the opportunity to ask questions and take as much time as required to decide if they would like to participate. In addition, once consent is obtained, subjects will undergo an initial screening treadmill run to ensure foot strike and cadence inclusion criteria are met.

Before the study begins, participants will be provided with a written consent form and be given the opportunity to ask any further questions. Prior to initiation of initial screening, data collection, or treatment, participants must sign the consent form.

Participants will be randomly assigned via computer to one of two treatment conditions: 1) increased cadence running gait or 2) forefoot strike running gait.

STUDY PROCEDURES

Subjects will have 13 visits to the Spaulding National Running Center for screening, interventions, and biomechanical analyses. Each visit is outlined below: Visit 1 (2.5 hours) determine if subject uses habitual heel strike and cadence less than or equal to 170, color vision test measure subject's weight, height, leg length, and arch height Baseline biomechanical analysis on instrumented treadmill Physical therapist-researcher will instruct strengthening exercises for feet and legs Subjects told to perform exercises daily and keep journal for 4 weeks

Visit 2 (30 minutes) One week after exercise instruction, subjects meet with a physical-therapist researcher to review and perform strengthening exercises and voice any questions or concerns

Visits 3-10 (1 hour each) Gait retraining on a treadmill using auditory feedback (metronome for cadence or Noraxon system for forefoot strike) and verbal instruction from a physical therapist.

These visits will be distributed over a 2-3 week time period. Subjects may run 2 days in a row, but never 3 days in a row.

Visit 11 (1 week after final gait retraining) (2 hours) Measure subject's resting heart rate, weight, height, leg length, and arch height Biomechanical analysis of running gait on instrumented treadmill Biomechanical analysis of running gait on instrumented treadmill until either 85-90 percent of age predicted heart rate is reached or a Borg Rating of Perceived Exertion score of greater than or equal to 17 is reached.

Subjects instructed in use of REDCap secure web application for journal of running frequency and distance (in miles), any discomfort or injuries that occur with running over the next 6 months.

Visit 12 (1 month after final gait retraining) (2 hours)

Measure subject's weight, height, leg length, and arch height Biomechanical analysis on instrumented treadmill Remind subjects to continue to keep journal

Reminder via email or phone call Physical therapist-researcher will contact subjects 1 time per month over the next 5 months to remind them to continue keeping journal of running frequency and distance (in miles), and any discomfort or injuries that occur.

Visit 13 (6 months after final gait retraining) (2 hours) Measure subject's weight, height, leg length, and arch height Biomechanical analysis on instrumented treadmill

The outcomes to be measured may include any combination of the following:

Structural measures: Height, weight, leg length, arch height. Video analysis: Digital video will only record the waist and below. Motion analysis: recording 3 dimensional movements using a computerized system with reflective markers attached to the body and high-speed cameras.

Ground reaction forces: gathered through force sensing platforms embedded in the treadmill Impact: an accelerometer attached to the body to record the impact experienced by the body with each footstrike.

Devices to be used The data will be collected using 3D motion capture (Vicon Motion Systems) in conjunction with 2 force plates (AMTI), which are embedded in the treadmill. Other devices to be used are foot calipers for arch height, a digital metronome, and an accelerometer with auditory feedback (Noraxon). These are all minimally invasive procedures that involve attaching sensors or markers to the skin and recording the output from the sensor.

d) Procedures/interventions All study procedures will take place at the Spaulding National Running Center in the Instrumented Treadmill Lab and clinic. Biomechanical Analysis

All biomechanical analyses of running gait will take place in the Treadmill Lab using an instrumented treadmill (AMTI) and a 3D motion analysis system. Four biomechanical analyses will be conducted over the duration of this investigation. These will occur at baseline, 1 week after the final gait retraining session, 1 month following gait retraining, and 6 months following gait retraining. Procedures for each analysis are as follows:

Subjects will run for a 3 minute warm up and be allowed to adjust to a speed of their preference. An investigator will control treadmill speed, but both participant and investigator can stop the treadmill at anytime via the emergency stop buttons. After warm up, data collection will occur for 4000 frames (15-20 steps). To minimize or prevent any laboratory performance effects, subjects will be distracted during data recording. The distraction technique is based on the Stroop Color and Word Test, and involves subjects reading aloud words on a screen directly in front of the treadmill. The correctness of the test is of no interest; rather, it only serves as a distraction technique.

Fatigue run One week after the final gait retraining session, subjects will be asked to run until they feel fatigued. Fatigue will be defined as either of the following two criteria: when the subject reaches 85-90 percent of age predicted heart rate max or when they report a score greater than or equal to 17 on the Borg Rating of Perceived Exertion scale. Once fatigue is reached, data will be collected for 4000 frames (15-20 steps).

Strengthening exercises During the first visit, a physical-therapist investigator will instruct subjects in strengthening exercises for the feet and legs. These activities will prepare musculoskeletal tissues to adapt to new forces they will experience during gait retraining. Subjects will be instructed to perform the exercises daily for 4 weeks, and will be given a journal to record their exercise performance. One week after exercise instruction, subjects will meet with the physical therapist-investigator to review the strengthening exercises and report any questions or concerns.

Gait Retraining

There will be 8 gait-retraining sessions over a 2-3 week time period. Subjects will be randomly assigned to either an increased cadence gait or a forefoot strike gait. The gait retraining protocols will be conducted on a treadmill (Woodway) in the clinic of the Spaulding National Running Center in the following manner:

Increased cadence (CAD) Protocol: After a 3-minute warm up, subjects' preferred step rate will be determined during their self-selected moderate intensity run for an additional 3 minutes using a visual count of footstrikes. Subjects will then be asked to increase their normal cadence by 7.5 percent while maintaining their speed. This will be accomplished by having subjects match their footstrikes to the beat of an audible digital metronome.

Forefoot strike (FFS) Protocol: Subjects will wear an accelerometer on the right anterior distal tibial. After a 3-minute warm up run, subjects will continue running for an additional 3 minutes and a baseline rearfoot strike accelerometer value will be recorded. Next, subjects will be instructed to land gently on the ball of their foot and lower their heels to the ground. They will be guided with verbal cues and visual inspection from a physical therapist. A forefoot strike accelerometer value will be recorded. If this value is exceeded, the device will provide audible feedback when a heel strike is detected signaling the runner to land with a FFS pattern.

For both groups, run time will be gradually increased from 10-30 minutes over 8 sessions. The auditory feedback will be provided constantly for the first 4 sessions and then gradually decreased in a systematic manner for the last four sessions. This feedback schedule has produced successful outcomes in a number of gait retraining studies.4,5,6 The feedback schedule for both groups is detailed as follows:

Session 1 - 10 minute treadmill run with metronome auditory feedback 100 percent of the time

Sessions 2,3,4 - Time of run will be gradually increased over sessions 2,3,4 to 12, 15, and 18 minutes respectively. Auditory feedback 100 percent of the time.

Sessions 5,6,7,8 - Time of run will be gradually increased over sessions 5,6,7,8 to 21,24,27, and 30 minutes respectively. Auditory feedback will be gradually reduced and given only at the beginning, middle, and end of a run.

This will be 4 minutes for sessions 5; 3 minutes for session 6; 2 minutes for session 7; and 1 minute for session 8.

Participants will be instructed not to run at any other time outside of the gait-retraining period. After completion of gait retraining, subjects will be encouraged to continue their new gait pattern as they run independently in the community. They will be instructed to increase running distance by no greater than 10 percent per week until they reach their desired running duration or distance. Subjects will be asked to keep journals of running activity after gait retraining until they return for the final gait analysis. This will be done via the REDCap (Research Electronic Data Capture) secure web application.

Data to be collected and when the data is to be collected:

Biomechanical outcomes as described above will be collected during each of the 5 biomechanical analyses that participants attend at the Spaulding National Running Center. Every effort will be made to accommodate participants' schedules for these sessions. Data collection will occur at the first visit (baseline), 1 week following gait retraining (approximately 7 to 8 weeks from baseline), 1 month after gait retraining (approximately 11 weeks from baseline), and 6 months after gait retraining (approximately 35 weeks from baseline).

Journals of daily strengthening exercise performance will be collected at Visit 3 (4 weeks from baseline). Journals of running frequency and distance and any discomfort or injuries will be collected throughout the 6 month follow up period using REDCap secure web application (9 to 35 weeks from baseline).

ELIGIBILITY:
Inclusion Criteria:

* history of running-related injury (outside of the past 3 months)
* ages 18 to 50 years
* currently running 5 to15 miles per week for at least 3 months
* habitual running cadence of less than or equal to 170 steps/min
* no contraindications for exercise as determined by the Physical Activity Readiness Questionnaire (PAR-Q).

Exclusion Criteria:

* do not use a heel strike as their habitual gait pattern
* habitual cadence greater than 170 steps/min
* history of injury within the past 3 months
* any history of stress fracture to any bone of the foot or ankle
* any past injuries or surgeries that have permanently altered gait
* color blindness

Injury will be defined as:

Running-related (training or competition) musculoskeletal pain in the lower limbs that causes a restriction on or stoppage of running (distance, speed, duration or training) for at least seven days or three consecutive scheduled training sessions, or that requires the runner to consult a physician or other health professional

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Vertical Load Rates | baseline, 1 week follow up, 1 month follow up, 6 month follow up
  average rate of loading calculated from Vertical Ground Reaction Force
Change in Foot Angle | baseline, 1 week follow up, 1 month follow up, 6 month follow up
  angle of foot in relation to ground, determines foot strike type
Change in running cadence (steps per minute) | baseline, 1 week follow up, 1 month follow up, 6 month follow up
  number of steps taken per minute

CONTACTS AND LOCATIONS:
Overall Officials: Irene Davis, PhD, Study Director — Director, Spaulding National Running Center

IPD SHARING:
Plan to Share IPD: No